CLINICAL TRIAL: NCT06039280
Title: Comparison of Dexamethasone and N Acetylcysteine (NAC) Versus N Acetylcysteine (NAC) Alone in the Prevention of Post Embolization Syndrome in Patients With Hepatocellular Carcinoma Following Transarterial Chemoembolization - Randomized Controlled Trial.
Brief Title: Comparison of Dexamethasone and N Acetylcysteine (NAC) Versus N Acetylcysteine (NAC) Alone in the Prevention of Post Embolization Syndrome in Patients With Hepatocellular Carcinoma Following Transarterial Chemoembolization.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HCC-06
Record Dates: First submitted 2023-08-04; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Acetylcysteine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC+Dexamethasone (Experimental): NAC started at 12 hr prior to procedure - (150 mg/kg/hr for 1 hr followed by 12.5 mg/Kg/hr for 4 hr, then continuous infusion of 6.25 mg/h for 48 after the procedure.
  Dexamethasone 20 mg in 5 ml NS 1 hour prior to procedure and 8 mg in 5 ml NS at day 2, day 3. Placebo 5 ml NS 1 hr prior to procedure.
  Interventions: Drug: N Acetylcysteine; Drug: Dexamethasone
- NAC+Placebo (Active Comparator): NAC started at 12 hr prior to procedure - (150 mg/kg/hr for 1 hr followed by 12.5 mg/Kg/hr for 4 hr, then continuous infusion of 6.25 mg/h for 48 after the procedure.
  Interventions: Drug: N Acetylcysteine; Other: Placebo

INTERVENTIONS:
Drug: N Acetylcysteine — NAC started at 12 hr prior to procedure - (150 mg/kg/hr for 1 hr followed by 12.5 mg/Kg/hr for 4 hr, then continuous infusion of 6.25 mg/h for 48 after the procedure.
Drug: Dexamethasone — Dexamethasone 20 mg in 5 ml NS 1 hour prior to procedure and 8 mg in 5 ml NS at day 2, day 3. Placebo 5 ml NS 1 hr prior to procedure.
  Arms: NAC+Dexamethasone
Other: Placebo — The placebo will be administered in the same way as the drug in the experimental group.
  Arms: NAC+Placebo

SUMMARY:
N-acetylcysteine (NAC), a glutathione precursor and potent antioxidant, is known as a liver protector. As a steroid preparation, dexamethasone is known to have efficient anti-inflammation and immunosuppression effects. N-acetyl cysteine and Dexamethasone's roles in preventing post-embolization syndrome following TACE have each been researched individually in the past. Up until now, no study has been done that has compared dexamethasone and NAC in post-embolization syndrome. With this study, we aim to study the efficacy of combining dexamethasone with N-acetyl cysteine in the prevention of post-embolization syndrome within 72 hours among patients who undergo transarterial chemoembolization for HCC.

DETAILED DESCRIPTION:
Aim & Objectives Hypothesis: The combination of dexamethasone with NAC is superior to NAC alone in prevention of PES among patients who undergo TACE in HCC as both medications work differently to prevent PES.

AIM:- To study the efficacy of combining Dexamethasone to N acetyl cysteine in prevention of post embolization syndrome within 72 hours among patients who undergo transarterial chemoembolization for HCC.

Objective - PRIMARY Prevention of post embolisation syndrome within 72 hours.

SECONDARY

* Prevention of post embolisation decompensation at 2 weeks.
* Decrease in the duration of hospitalization.
* To study the adverse effects of NAC and steroids in patients who undergo transarterial chemoembolisation for HCC.

Methodology:

Study population:

* All patients undergoing TACE procedure
* Valid Consent
* Age 18-65 years

Study design:

Monocentric open label prospective randomized controlled study. The study will be conducted in Department of Hepatology, ILBS.

Sample size:

* Assuming that NAC prevents PES by 75% and addition of dexamethasone further prevents PES by 20 % (i.e combination of NAC and Dexamethasone prevents total 95%).
* Then with alpha as 5% and power 90 % .we need to enroll total 130 cases i.e 65 in each arm.
* Further assuming 10% drop out , it is decided to enroll 150 cases i.e. 75 in each arm.
* Allocation will be done randomly by block randomization method, taking block size as 10.

Monitoring and assessment: All the parameters of the objective and also noted any adverse effects.

Intervention: TACE.

STATISTICAL ANALYSIS:

The data will be entered in Microsoft excel and will be analyzed using SPSS version 22. The categorical data will be analyzed using Chi square/Fissure test. Exact test and continuous data will be compiled using t-test. Besides this the univariate and multivariate survival analysis will be carried out using Cox regression method. Kaplan-Meier technique will be applied for further analysis. P-value<0.05 will be considered as significant.

Adverse effects: allergic drug reaction.

Stopping rule: If patient decided to withdraw from study.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing TACE procedure
* Valid Consent
* Age 18-65 years

Exclusion Criteria:

* Child Pugh C, Child Pugh B > 8
* HCC patients with a curative therapy (Ablation, Resection or LT)
* ECOG Performance Status 3-4
* Pregnancy
* History of allergic reaction from NAC
* significant cardiopulmonary disease
* UGI bleed within last 28 days
* Recent surgery within last 28 days
* Documented febrile illness in last 1 weeks
* Uncontrolled Diabetes (FBS > 200, HBA1C > 8)
* Uncontrolled Hypertension (BP > 160/100)
* Structural kidney disease with eGFR < 60 ml/min

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Prevention of post-embolization syndrome | 72 hours
  Prevention of Post-embolization syndrome , Defined base on South west oncology group (SWOG) toxic coding less than 2 score

SECONDARY OUTCOMES:
Prevention of post TACE decompensation at 4 weeks | 4 weeks
  Metric / Method of measurement : Post TACE decompensation defined as an increase in Child-Pugh score of more than two points or newly developed decompensating events, such as ascites, hepatic encephalopathy, or serum total bilirubin > 2 mg/dL.
Decrease in the duration of hospitalisation | 4 weeks
Adverse events of Dexamethasone and NAC in patients undergoing transarterial chemoembolisation for HCC | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No